CLINICAL TRIAL: NCT04045626
Title: Study of Demarcation Line Depth in Transepithelial Versus Epithelium-off Accelerated Cross-linking (AXL) in Keratocouns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Sarah Akram Azzam, Principal investigator, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N28
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Progressive Keratoconus
MeSH Terms: interventions — Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transepithelial accelerated cross-linking (Active Comparator): Paracel is instilled 1 drop every 1.5 minutes for 4.5 minutes then vibex-xtra is instilled 4 drops at 5.5 minutes followed by 1 drop at 6.5 minutes for a total soak time of 11 minutes followed by ultraviolet-A" UVA" irradiation with intended irradiance of 45mW/cm2 for 2.4 minutes
  Interventions: Procedure: corneal cross-linking
- Epithelium-off accelerated cross-linking (Active Comparator): Vibex-rapid is instilled every 2 minutes for 10 minutes followed by ultraviolet-A "UVA" irradiation of 30 mW/cm2 for 4 minutes
  Interventions: Procedure: corneal cross-linking

INTERVENTIONS:
Procedure: corneal cross-linking — Riboflavin is instilled over cornea followed by Ultraviolet-A irradiation

SUMMARY:
To assess depth of demarcation line in transepithelial versus epithelium-off accelerated cross-linking in keratoconus patients

DETAILED DESCRIPTION:
Anterior segment optical coherence tomography "OCT" will be performed to evaluate the corneal stroma for the presence of demarcation line 1 month postoperatively by an independent observer unware of purpose of study

ELIGIBILITY:
Inclusion Criteria:

* progressive keratoconus stage 1-2

Exclusion Criteria:

* any concomitant ocular disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
evaluation of depth of demarcation line | 1 month postoperative
  Anterior segment optical coherence tomography "AS-OCT" is used to measure depth of demarcation line

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Azzam, MD, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- Kasr Al Ainy teaching hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salah Y, Omar K, Sherif A, Azzam S. Study of Demarcation Line Depth in Transepithelial versus Epithelium-Off Accelerated Cross-Linking (AXL) in Keratoconus. J Ophthalmol. 2019 Sep 26;2019:3904565. doi: 10.1155/2019/3904565. eCollection 2019. PMID 31662893